CLINICAL TRIAL: NCT01944332
Title: Gamete Treatment to Correct Fertilization Failure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0712009553
Record Dates: First submitted 2013-07-08; First posted 2013-09-17 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Infertility
Keywords: gamete treatment; ICSI; IVF; infertility; oocyte activation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gamete treatment- oocytes and sperm (Experimental): The spermatozoa will be prepared in the standard fashion and utilized for injection after exposure to a membrane permeabilizing agent. Patient specimen will be selected through a synthetic, sterile, single-use, culture-tested mesh. The specimen will then be placed in a 37°C environment. After 30 minutes, the selected portion is retrieved from the other side of the mesh. The injected oocytes will be then exposed to the previously mentioned activating agents for the purpose of inducing embryo development. The successfully fertilized oocytes will be further kept in culture for up to 5 days as per standard IVF/ICSI.
  Interventions: Procedure: gamete treatment

INTERVENTIONS:
Procedure: gamete treatment — Patient specimen will be selected through a synthetic, sterile, single-use, culture-tested mesh. The specimen will then be placed in a 37°C environment. After 30 minutes, the selected portion is retrieved from the other side of the mesh. The spermatozoa will be prepared in the standard fashion and utilized for injection or intrauterine insemination after exposure to a membrane permeabilizing agent. Human recombinant PLC-zeta will also be used if the spermatozoa have been confirmed to be PLC-zeta deficient. The injected oocytes will then be exposed to activating agents for the purpose of inducing embryo development. The oocyte activating agent is calcium ionophore and for sperm membrane permeabilization to assist in sperm DNA decondensation is streptolysin O (SLO).

SUMMARY:
In this proposed research study, the investigators plan to assess the efficacy of gametes' (egg and sperm) treatment on fertilization as well as pre- and post-implantation embryo development.

DETAILED DESCRIPTION:
The spermatozoa will be prepared in the standard fashion and utilized for injection after exposure to a membrane permeabilizing agent. The raw sperm specimen may be selected through a synthetic, sterile, single-use, culture-tested mesh. The specimen will then be placed in a 37°C environment. After 30 minutes, the selected portion is retrieved from the other side of the mesh. The spermatozoa will be prepared in the standard fashion will be utilized for injection or intrauterine insemination. Human recombinant PLC-zeta will also be used if the spermatozoa have been confirmed to be PLC-zeta deficient.

The injected oocytes will be then exposed to the previously mentioned activating agents for the purpose of inducing embryo development. The successfully fertilized oocytes will be further kept in culture for up to 5 days as per standard IVF/ICSI. Results in terms of fertilization and embryo cleavage will be assessed and monitored for the remainder of the culture period. Developing embryos selected according to standard criteria will be replaced to the patient or will be cryopreserved.

Because fertilization failure carries such a high emotional and financial toll on our patients, at the present time, the only method to generate an embryo for these cases is to perform assisted oocyte activation in conjunction with ICSI. The research intervention - assisted oocyte activation - is believed to help alleviate the failed fertilization by obtaining some zygotes for the patient. In these cases of complete failed fertilization, intracytoplasmic sperm injection (ICSI) will be performed as a routine clinical treatment even if they are not enrolled in the study. After several failures, their reproductive physician may recommend the use of donor spermatozoa instead of the male partner's.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete fertilization failure with standard IVF or failure with one prior ICSI treatment cycle

Exclusion Criteria:

* not meeting inclusion criteria
* IVF without ICSI

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2007-09 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Fertilization rate | 2 months
  Efficacy of gamete treatment on fertilization

CONTACTS AND LOCATIONS:
Overall Officials: Gianpiero Palermo, MD, MPH, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Center fo Reproductive Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No